CLINICAL TRIAL: NCT03501173
Title: A Multicentre Cohort Study of Patients With Advanced Prostate Cancer in Canada
Brief Title: A Study of Participants With Advanced Prostate Cancer in Canada
Acronym: GURC
Status: Completed | Type: Observational
Sponsor: Janssen Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108454; 212082PCR4049 (Other: Janssen Inc.)
Record Dates: First submitted 2018-03-28; First posted 2018-04-18 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Metastatic Castrate-Sensitive Prostate Cancer (mCSPC): Participants will be defined as having mCSPC if there is a new mCSPC diagnosis in the past 6 months, documented metastatic prostate cancer, no more than 12 months of androgen deprivation therapy (ADT) in any setting and no more than 6 months of systemic treatment for mCSPC (example, next generation androgen receptor targeted therapy or chemotherapy).
  Interventions: Other: Standard of Care
- Metastatic Castrate-Resistant Prostate Cancer (mCRPC): Participants will be defined as having mCRPC if there is mCRPC diagnosis at any time, documented metastatic prostate cancer, documented castration resistance per Prostate Cancer Working Group 2 criteria (elevated prostate specific antigen [PSA] despite testosterone less than [<]50 nanogram per deciliter [ng/dL] [<1.7 nano moles per liter{nmol/L}]), the first treatment for mCRPC was started in the past 6 months or is scheduled to begin.
  Interventions: Other: Standard of Care
- NonMetastatic Castrate-Resistant Prostate Cancer (nmCRPC): Participants will be defined as having nmCRPC if there is nmCRPC diagnosis at any time, documented non-metastatic prostate cancer, documented castration resistance per Prostate Cancer Working Group 3 criteria (elevated PSA despite testosterone <50 ng/dL [<1.7 nmol/L]). nmCRPC, defined as a prostate specific antigen doubling time (PSADT) of less than or equal to 12 months, or beginning next generation ARAT for nmCRPC.
  Interventions: Other: Standard of Care
- mCRPC (Treatment-experienced in the nmCRPC or mCSPC Setting): Participants will be defined as having mCRPC (treatment-experienced in the nmCRPC or mCSPC setting) if there is nmCRPC diagnosis at any time, documented non-metastatic prostate cancer, documented metastatic prostate cancer, documented castration resistance per Prostate Cancer Working Group 2 criteria (elevated PSA despite testosterone <50 ng/dL [<1.7nmol/L]), the first treatment for mCRPC clinical state was started in the past 6months or is scheduled to begin, disease progression occurred while receiving active treatment (ARAT or chemotherapy) in the prior nmCRPC or mCSPC clinical state.

INTERVENTIONS:
Other: Standard of Care — Participants will not receive any intervention in this study. Participants will receive standard of care therapy.
  Groups: Metastatic Castrate-Resistant Prostate Cancer (mCRPC); Metastatic Castrate-Sensitive Prostate Cancer (mCSPC); NonMetastatic Castrate-Resistant Prostate Cancer (nmCRPC)

SUMMARY:
The purpose of this study is to document the course of advanced prostate cancer in Canada in terms of disease progression, real-world treatment, and patient management.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a confirmed diagnosis of adenocarcinoma of the prostate
* Participant must have prostate cancer, as follows: a) nonmetastatic castrate-resistant prostate cancer (nmCRPC): nmCRPC diagnosis at any time; documented castration resistance per Prostate Cancer Working Group 3 criteria23 (elevated prostate specific antigen [PSA] despite testosterone less than (<) 50 nanograms per deciliter [ng/dL] [<1.7 nano moles per liter {nmol/L}]); Negative for metastases on conventional imaging (computerized tomography, Magnetic resonance imaging, bone scans); Prostate specific antigen doubling time (PSADT) less than equal to (<=) 12 months within the last 6 months or beginning treatment with approved next-generation ARAT for treatment of nmCRPC; b) Metastatic castrate-sensitive prostate cancer (mCSPC): new mCSPC diagnosis in the past 6 months (can be de novo or primary progressive recurrent following local radical therapy); documented metastatic prostate cancer; no more than 12 months of androgen deprivation therapy (ADT) in any setting; no more than 6 months of systemic treatment for mCSPC (example, approved next generation androgen receptor targeted therapy or chemotherapy]); c) Metastatic castrate-resistant prostate cancer (mCRPC): mCRPC diagnosis at any time; documented metastatic prostate cancer; documented castration resistance per Prostate Cancer Working Group 2 criteria (elevated prostate specific antigen [PSA] despite testosterone less than [<]50 nanogram per deciliter [ng/dL] [<1.7 nmol/L]); the first treatment for mCRPC was started in the past 6 months or is scheduled to begin; d) mCRPC (treatment-experienced in the nmCRPC or mCSPC setting): mCRPC diagnosis at any time; documented metastatic prostate cancer; documented castration resistance per Prostate Cancer Working Group 2 criteria (elevated PSA despite testosterone <50 ng/dL [<1.7 nmol/L]); the first treatment for mCRPC clinical state was started in the past 6 months or is scheduled to begin; disease progression occurred while receiving active treatment (androgen receptor-axis therapy [ARAT] or chemotherapy) in the prior nmCRPC or mCSPC clinical state
* Participant must have a life expectancy of more than 6 months
* Participant must sign (and/or their legally acceptable representative, if applicable) a participation agreement/informed consent form (ICF) allowing data collection and source data verification in accordance with local requirements and/or sponsor policy

Exclusion Criteria:

* At the time of screening, patient is currently enrolled in other Janssen sponsored clinical study (any indication) or an interventional clinical trial investigating a non Health Canada approved drug and/or procedure for the treatment and/or monitoring of prostate cancer (Janssen or non-Janssen company sponsored)
* Participant is currently enrolled in any observational study sponsored or managed by a Janssen company

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant having advanced prostate cancer (metastatic castrate-sensitive prostate cancer [mCSPC] or metastatic castrate-resistant prostate cancer [mCRPC] or nonmetastatic castrate-resistant prostate cancer [nmCRPC]) or mCRPC (treatment-experienced in the nmCRPC or mCSPC setting) will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Time to Prostate Specific Antigen (PSA) Progression | Approximately up to 5 years
  Time to PSA progression is defined as the time interval from the date of start of study enrollment to the date of first evidence of PSA progression. In participants whose PSA level has decreased, PSA progression is defined as at least a 25 percent (%) increase from nadir (lowest value including the most recent value prior to study enrollment) and an increase in the absolute value of 2 nanogram per milliliter (ng/mL) or greater, confirmed by a subsequent measurement at least 3 weeks after the increase. In participants whose PSA level has not decreased, PSA progression is defined as at least a 25% increase from the most recent value prior to study enrollment and an increase in the absolute value of 2 ng/mL or greater after 12 weeks.
Time to Radiographic Evidence of Disease Progression | Approximately up to 5 years
  Time to radiographic evidence of disease progression is defined as the time interval from the date of start of study treatment to the date of first appearance of 2 or more new bone lesions on bone scan or enlargement of a soft tissue lesion using the Response Evaluation Criteria in Solid Tumors (RECIST).
Time to Skeletal-Related Events | Approximately up to 5 years
  Time to skeletal-related events is defined as the time interval from the date of start of study treatment to the date of first skeletal-related event.
Time to Death | Approximately up to 5 years
  Time to death is defined as the time interval from the date of start of study enrollment to death.
Number of Participants with Different Primary Causes of Death | Approximately up to 5 years
  The number of participants with different primary causes of death will be reported.
Time to Progression from mCSPC to mCRPC in Participants with mCSPC | Approximately up to 5 years
  In participants with mCSPC, time to progression from mCSPC to mCRPC is defined as the time interval which is either calculated from date when mCSPC was first documented or from the date of start of study treatment, if participant receives treatment for mCSPC to the progression to mCRPC.
Time from Biochemical Recurrence (BCR) to Nonmetastatic Castrate-Resistant Prostate Cancer (nmCRPC) and nmCRPC to mCRPC | Approximately up to 5 years
  In participants with mCRPC, time from BCR to nmCRPC and nmCRPC to mCRPC will be analyzed retrospectively. BCR is defined as PSA greater than (>)0.2 nanogram per milliliter (ng/mL) after radical prostatectomy and PSA >2 ng/mL above the nadir (lowest value including the most recent value prior to study enrollment) after radical radiotherapy.
Number of Participants with PSA Testing from BCR to nmCRPC and nmCRPC to mCRPC, in Participants with mCRPC | Approximately up to 5 years
  In participants with mCRPC, number of participants having PSA testing from BCR to nmCRPC and nmCRPC to mCRPC will be reported.
Number of Participants with Frequency of Imaging from Time of BCR to nmCRPC and nmCRPC to mCRPC | Approximately up to 5 years
  In participants with non metastatic castrateresistant prostate cancer (nmCRPC), number of participants having imaging from BCR to nmCRPC and mCRPC to nmCRPC will be reported.
PSA Level at Start of Androgen Deprivation Therapy (ADT) in Participants with mCRPC | Approximately up to 5 years
  In participants with mCRPC, PSA level at start of ADT will be reported.
PSA Doubling Time (PSADT) at the Detection of Castration Resistance in Participants with mCRPC | Approximately up to 5 years
  In participants with mCRPC, PSADT at the detection of castration resistance will be reported. PSADT is the length of time it takes for a PSA to double based on an exponential growth pattern.
Time from nmCRPC to High-Risk (HR) nmCRPC | Approximately up to 5 years
  Time from nmCRPC to HR nmCRPC is defined as prostate specific antigen doubling time (PSADT) less than or equal to (<=) 10 months.
Time from ADT Initiation to nmCRPC | Approximately up to 5 years
  Time from ADT initiation to nmCRPC will be reported.
Median Absolute prostate specific antigen (PSA) at onset of HR-nmCRPC | Approximately up to 5 years
  Median absolute PSA at onset of HR-nmCRPC will be reported.
Time to Initiation of Subsequent Prostate Cancer Treatment | Approximately up to 5 years
  Time to initiation of subsequent prostate cancer treatment is defined as the time interval from the date of start of study treatment to the date of start of subsequent prostate cancer treatment.
Duration of Each Therapy | Approximately up to 5 years
  Duration for each therapy will be reported for all participants.
Percentage of Participants Receiving Chemotherapy, Other Drug Treatments, or no Drug Treatment | Approximately up to 5 years
  Percentage of participants receiving chemotherapy, other drug treatments, or no drug treatment, will be reported for all participants.
Time to Treatment Initiation | Approximately up to 5 years
  Time to treatment initiation, will be reported for all participants.
Time to Dose Modification | Approximately up to 5 years
  Time to dose modification, will be reported for all participants.
Number of Participants who Switch the Treatment | Approximately up to 5 years
  Number of participants who switch the treatment, will be reported.
Number of Participants who Discontinued the Treatment | Approximately up to 5 years
  Number of participants who discontinued the treatment, will be reported.
Most Common Sequences for Lines of Therapy in Participants with mCRPC | Approximately up to 5 years
  In participants with mCRPC, most common sequences for lines of therapy will be reported.
Number of Participants Retreated with Docetaxel in Participants with mCRPC | Approximately up to 5 years
  In participants with mCRPC, number of participants having retreatment with docetaxel will be reported.
Percentage of Participant with Radiographic Imaging Modality | Approximately up to 5 years
  Percentage of participants with radiographic imaging modality which includes bone scan, magnetic resonance imaging, ultrasound, X-ray will be reported.
Number of Days Hospitalized for Prostate Cancer or Treatment of Prostate Cancer | Approximately up to 5 years
  Number of days for which participant was hospitalized for prostate cancer or treatment of prostate cancer, will be reported for all participants.
Number of Visits to Emergency Department for Prostate Cancer or Treatment of Prostate Cancer | Approximately up to 5 years
  Number of visits to emergency department for prostate cancer or treatment of prostate cancer, will be reported for all participants.
Number of Outpatient Visits to Specialists Involved in Management of Prostate Cancer | Approximately up to 5 years
  Number of outpatient visits to specialists (urologist, medical oncologist, uro-oncologist, radiation oncologist) involved in management of prostate cancer, will be reported for all participants.
Dates of Genomic or Genetic Testing | Approximately up to 5 years
  Dates of genomic or genetic testing (including dopa-responsive dystonia [DRD]/ homologous recombination repair [HRR]/ breast cancer gene-1 [BRCA1]/ BRCA2/ataxia-telangiesctasia mutated [ATM]/partner and localizer of the BRCA2 gene [PALB2]/ androgen receptor [AR]) will be reported.
Types of Genomic or Genetic Testing | Approximately up to 5 years
  Types of genomic or genetic testing (including DRD/HRR/ BRCA1/ BRCA2/ATM /PALB2/AR) will be reported.
Charlson Comorbidity Index Score | Approximately up to 5 years
  Charlson Comorbidity Index score will be summarized descriptively. The Charlson Comorbidity Index is a 19-item measure assessing comorbid conditions. The total possible score on the Charlson Comorbidity Index ranges from 0 to 37. If a condition is not present, the score for that condition is zero. The higher scores indicate greater comorbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Inc. Clinical Trial, Study Director — Janssen Inc.
Locations (22):
- Canada (22):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Prostate Cancer Centre, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Abbotsford Regional Hospital and Cancer Centre BC Cancer Agency, Abbotsford, British Columbia
  - British Columbia Cancer Agency(BCCA)-Sindi Ahluwalia Hawkins Centre for the Southern Interior(CSI), Kelowna, British Columbia
  - Vancouver General Hospital / Vancouver Prostate Centre, Vancouver, British Columbia
  - BC Cancer Agency - Vancouver BC, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II - Health Sciences Centre, Halifax, Nova Scotia
  - G. Kenneth Jansz Medicine, Burlington, Ontario
  - Research St. Joseph's - Hamilton, Hamilton, Ontario
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Lawson Health Research Institute, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Scarborough Health Network, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Urology South Shore Research, Greenfield Park, Quebec
  - CHUM - Centre hospitalier universitaire de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Québec Université Laval, Québec, Quebec